CLINICAL TRIAL: NCT01076335
Title: Phase II Study of Neoadjuvant Hormonal Therapy Plus Docetaxel Followed by Radical Prostatectomy for Men With Proven or Suspected Node-positive Prostate Cancer
Brief Title: Neoadjuvant Hormones + Docetaxel in Node-Positive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0273; P50CA090270 (NIH); NCI-2010-01369 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
Keywords: Neoadjuvant Hormonal Therapy; Docetaxel; Taxotere; Chemotherapy; Radical Prostatectomy; Node-positive Prostate Cancer; Androgen-dependent prostate cancer; Lymph node metastases
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis | interventions — Leuprolide; Goserelin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Hormones + Docetaxel (Experimental): Neoadjuvant Hormonal Therapy plus Docetaxel followed by Radical Prostatectomy
  Interventions: Drug: Neoadjuvant Hormonal Therapy; Drug: Docetaxel

INTERVENTIONS:
Drug: Neoadjuvant Hormonal Therapy — Monthly or quarterly LHRH Agonist Depot injection (leuprolide or goserelin acetate) for one year.
  Other Names: Leuprolide Acetate; Goserelin Acetate
Drug: Docetaxel — 35 mg/m2 by vein (IV) on Day 1, 8, 15 and 22 every 6 weeks.
  Other Names: Taxotere

SUMMARY:
The goal of this clinical research study is to find out if a therapy using docetaxel chemotherapy with hormonal therapy taken before your scheduled surgery is beneficial to treatment of prostate cancer. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Advanced prostate cancer may be responsive to a combination of hormonal and chemotherapy treatments. Researchers believe that the use of chemotherapy and hormonal therapy before your scheduled surgery may help to affect or delay the progression of prostate cancer.

Before surgery, you will have imaging studies, including a chest x-ray, CT scan and a bone scan. You may also have an MRI scan. These tests are being done to check on the status of the disease. You will also have 3 tablespoons of blood drawn for routine blood tests, before treatment.

All treatment will be given on an outpatient basis. Treatment should start as soon as possible, within 14 days after registration. You will receive hormonal treatment once a month for the 12 months before your surgery. Hormonal treatments will not continue after the surgery.

You will be given dexamethasone, Benadryl® (diphenylhydramine) and Pepcid® (famotidine) , by a vein in your arm or by central line in a vein before your therapy begins with docetaxel on Day 1 of the first treatment cycle. Dexamethasone will help decrease bone marrow inflammation. Diphenhydramine helps prevent allergic reactions. Famotidine protects you against stomach irritation by decreasing the amount of acid in your stomach.

Docetaxel will be given through a needle in your vein (IV) once a week during the first 4 weeks of each 6-week period (called a study cycle). Each dose of docetaxel will take about an hour to be given. The total treatment time to complete the docetaxel will be 3 study cycles (18 weeks). Before each 6-week study cycle with docetaxel, you will come to the clinic for a physical exam and routine blood tests (2 tablespoons).

After your treatment with docetaxel and hormones, you will then have an operation to remove the prostate gland and the tumor. Your doctor will discuss the surgical procedure with you in detail and explain the risks of the operation. You will need to sign a separate consent form before undergoing the surgical procedure.

After surgery, you will be closely checked for any possible side effects. After completion of the treatment, you will be monitored every 3 months for the first year and every 6 months for the second year. You will also have 2 tablespoons of blood drawn for routine blood test monitoring at every follow-up visit.

This is an investigational study. Docetaxel and the hormone treatments used in this study are FDA approved medications for the treatment of prostate cancer. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with adenocarcinoma of the prostate that in the opinion of the surgeon could be resectable after response to systemic therapy. Ductal carcinoma variant is included.
2. All patients must be regarded as acceptable anesthetic risk for radical prostatectomy and confirm their intention to undergo radical prostatectomy at the end of the neoadjuvant therapy.
3. Zubrod performance status 2 or better.
4. All patients must have thorough tumor staging and meet one of the following criteria: a) Either lymph node biopsy or lymph node dissection demonstrating presence of lymph node metastasis. b) Pelvic or retroperitoneal lymphadenopathy >/= 2.0 cm visualized on CT scan (biopsy is not required if >/= 2.0 cm and in typical distribution) c) Primary tumor Gleason score >/= 8 and serum PSA concentration >/= 25 ng/ml, indicating high risk of occult lymph node metastases.
5. (# 4 cont'd) d) Primary tumor stage T3 and Gleason score >/= 7, indicating high risk of occult lymph node metastases. e) Primary tumor stage T4 indicating high risk of occult lymph node metastases.
6. Prior hormonal therapy up to 6 months is permitted. No concurrent ketoconazole is permitted.
7. Patients must have adequate bone marrow function defined as an absolute peripheral granulocyte count of > 1,500/mm^3 and platelet count of > 100,000/mm^3; adequate hepatic function defined with a total bilirubin of < 1.5 mg/dl and AST/ALT < 2X the upper limits of normal; adequate renal function defined as serum creatinine clearance > 40 cc/min (measured or calculated).
8. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution.
9. All patients must be evaluated in the Department of Urology and Department of Genitourinary Medical Oncology prior to signing informed consent.

Exclusion Criteria:

1. Patients with small cell or sarcomatoid histology.
2. Patients with clinical or radiological evidence of bone or other extranodal metastasis (M1b or M1c).
3. Prior chemotherapy.
4. Patients with severe or uncontrolled intercurrent infection.
5. Patients with New York Heart Association (NYHA) Class III/IV congestive heart failure, unstable angina or history of myocardial infarction within the last 6 months.
6. Contraindications to corticosteroids.
7. Uncontrolled severe hypertension, persistently uncontrolled diabetes mellitus, oxygen-dependent lung disease, chronic liver disease or HIV infection.
8. Second malignancies (excluding non-melanoma skin cancer) unless disease-free for 3 years.
9. Overt psychosis, mental disability or otherwise incompetent to give informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Pagliaro, MD, BA, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: Enrollment took place from 21 April 2005 to 31 March 2008. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 40 enrolled, one participant (2.5%) declined presurgical therapy after enrollment and was excluded from subsequent analyses.
Groups:
- Neoadjuvant Hormones + Docetaxel: One year Neoadjuvant Hormonal Therapy of LHRH Agonist Depot injection (monthly or quarterly) plus three cycles Docetaxel 35 mg/m^2 weekly intravenous (IV) (approximately 4 months) followed by Radical Prostatectomy
Period: Overall Study
Arm/Group | Neoadjuvant Hormones + Docetaxel
Started | 40
Completed | 36
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Withdrawal without treatment | 1

BASELINE CHARACTERISTICS:
Population: One participant declined presurgical therapy after enrollment and was excluded from analysis.
Arm/Group | Neoadjuvant Hormones + Docetaxel
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 61.5 [38 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Progression Free at 1 Year
Description: Participants prostatic specific antigen (PSA) progression-free or event-free survival (that is, freedom from treatment failure) 1 year postoperatively. Treatment failure defined as objective tumor progression during therapy or in year after surgery, confirmed postoperative PSA ⩾1 ngml - 1, or any postoperative radiation, hormonal or other systemic therapy. Participants who did not undergo surgery within 8 weeks of completing 1 year of therapy on protocol (for any reason, including participant refusal) were counted as treatment failure, as were participants whose surgery was begun and aborted.
Time Frame: 1 Year
Population: One participant of 40 enrolled declined presurgical therapy after enrollment and was excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Hormones + Docetaxel
Number analyzed (Participants) | 39
participants | 13

ADVERSE EVENTS:
Time Frame: Adverse events collected through chemotherapy treatment and surgery, up to 18 weeks. One participant declined presurgical therapy after enrollment and was excluded from analysis.
Description: All toxicities encountered evaluated according to grading system (0-4) in NCI Common Toxicity Criteria v3.0 and recorded prior to each course of therapy along with duration and treatment. Surgical complications assessed during and within 90 days of procedure by using Clavien grading.
Arm/Group | Neoadjuvant Hormones + Docetaxel
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 39/39
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Hormones + Docetaxel (N=39)
Pericardial effusion (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) elevation (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema: limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (6)
Gastrointestinal-Other (Specity) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Hemoglobin decrease (Investigations) | 5 (5)
Hemorrhage pulmonary/upper respiratory(Nose) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Leukocytes Low (Total White Blood Count) (Investigations) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration--Depression (Psychiatric disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (General disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Ocular/Visual-Other (Eye disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 2 (2)
Uric acid, serum-high (hyperuricemia) (Renal and urinary disorders) | 1 (1)
Watery eye (epiphora, tearing) (Eye disorders) | 3 (3)
Weight loss (Investigations) | 2 (2)
Bladder spasms (Renal and urinary disorders) | 1 (1)
Superficial wound infection (Infections and infestations) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Anastomotic urine leak (Injury, poisoning and procedural complications) | 2 (2)
Pelvic lymphocele (Vascular disorders) | 1 (1)
Anastomotic stricture (Injury, poisoning and procedural complications) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes